CLINICAL TRIAL: NCT05503836
Title: Assessment of Different Scores for Prediction of Morbidity and Mortality in Cirrhotic Patients Undergoing Abdominal Surgeries
Brief Title: Assessment of Severity of Liver Disease Before Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tasneem Khaled, Assistant lecturer, Assiut University
Other Study IDs: surgery in cirrhotic patients
Record Dates: First submitted 2022-08-06; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: abdominal surgeries — abdominal surgeries

SUMMARY:
* Determine the ability of Child Pugh, MELD, and ALBI scores to predict mortality and morbidity in cirrhotic patients undergoing abdominal surgeries.
* Evaluate the prognostic efficacy of ALBI score versus CTP and MELD scores to predict mortality and morbidity in cirrhotic patients undergoing abdominal surgeries

DETAILED DESCRIPTION:
Cirrhotic patients have a great risk for increased morbidity and mortality rather than the normal population after undergoing surgical procedures.(1) High mortality rates were reported among patients with liver cirrhosis as high as 67 % after surgical interventions. (2) This high surgical risk occurs is contributing to the pathophysiology of the diseased liver itself and to the presence of contributing factors, such as coagulopathy, poor nutritional status, adaptive immune dysfunction, cirrhotic cardiomyopathy, and renal and pulmonary dysfunction, which all predisposing to poor outcomes. Preoperative optimization after risk stratification and careful management are mandatory before surgery.(1) The challenge is to assess the surgical risks before deciding whether the procedure will be carried out safely or should be delayed until the patient underwent liver transplantation, or it should be avoided completely, and so early involvement of an experienced surgical and medical team is important.(1) The degree of hepatic dysfunction is one of the most risk factors for post-operative mortality and complication, other factors are considered as non-hepatic comorbidities, type of surgical procedures and the expertise of the managing team.(3) Various score systems are being used in clinical practice, for assessment of prognosis among cirrhotic patients such as the Child-Turcotte score, Model for End stage Liver Disease (MELD), . However, these scoring systems have several limitations in their prognostic implications. Although CTP scoring is easily applicable at bedside, the interpretation of ascites and encephalopathy is subjective in nature and equal point allocation of all variables make its results unstable.(4, 5) Also, the wide reference ranges for grading cirrhosis and its complications, such as ascites, bleeding, spontaneous bacterial peritonitis (SBP), and hepato-pulmonary syndrome, restricts the predictive accuracy of the MELD score. This raises a need for evaluating other potential biomarkers to strengthen prognostication and severity of cirrhosis (3).

Recently, the albumin-to-bilirubin (ALBI) score has emerged to evaluate severity of liver disease in hepatocellular carcinoma (HCC) (5) The ALBI is a new and simple score, easily calculated at bedside without having to use subjective determinants such as ascites and encephalopathy and because the ALB and TB levels are indicators of liver function, and can reflect the synthesis and metabolic function of the liver , so Its prognostic role in various liver diseases has recently been validated in several studies where it was found to be superior to CTP and MELD in assessing severity of liver disease.(4, 6, 7)

In general, ALBI grades 1, 2, and 3 correspond to Child-Pugh A, B, and C, respectively, and it was reported that the ALBI grade is more accurate in prediction of postoperative liver failure than the Child-Pugh grade. However, the Child-Pugh grade itself is a relatively rough grading system and was not intended for the prediction of liver failure after hepatectomy .(8)

ELIGIBILITY:
Inclusion Criteria:

* o All confirmed cases of cirrhosis aged ≥ 18 years of either sex, admitted to the Assiut university hospitals for abdominal surgeries (elective or emergency) were enrolled in the study.

  * Cirrhosis is confirmed by the following diagnostic criteria :

    1. Clinical history and examination with special stress on symptoms and signs of chronic liver disease with or without evidence of hepatic decompensation e.g. the presence of ascites and with or without evidence of complications e.g. jaundice, bleeding varices, ascites, and lower limb edema.
    2. Laboratory findings in the form of raised bilirubin, impaired coagulation profile, and/or low serum albumin.
    3. Abdominal ultrasonography revealing liver cirrhosis (coarse echo pattern, attenuated hepatic veins, irregular outlines, hypertrophy of caudate lobe and/or shrunken liver, and presence of splenomegaly, ascites )

Exclusion Criteria:

* o Cirrhotic patients undergoing extra abdominal surgeries.

  * Patients admitted for liver transplantation.
  * Patients less than 18 years of age.
  * Patients refused to participate.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All confirmed cases of cirrhosis aged ≥ 18 years of either sex, admitted to the Assiut university hospitals for abdominal surgeries (elective or emergency) .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
frequency of deaths and number of cases with hepatic decompensation and compliication | Between August 2022 and August 2024
  As we will follow up the patient for 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: .Mohamed Omar, Professor, Study Director — Assiut University

REFERENCES:
- [Background] Naqvi IH, Talib A, Mahmood K, Abidi R, Rizvi SNZ. The ability of the new ALBI scoring in predicting mortality, complications and prognostic comparison among cirrhotics. Prz Gastroenterol. 2019;14(4):250-257. doi: 10.5114/pg.2019.83872. Epub 2019 Mar 25. PMID 31988671